CLINICAL TRIAL: NCT04155138
Title: Recipients With Limited Bimodal Benefit: HA or CROS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CRRF 842
Record Dates: First submitted 2018-10-18; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Cochlear Implant; Hearing Disability; Hearing Disorders and Deafness
Keywords: cochlear implant; hearing aid; cros device; bimodal
MeSH Terms: conditions — Hearing Disorders; Deafness

STUDY DESIGN:
Intervention Model Description: Naida Hearing Aid Naida CROS Device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naida Hearing Aid (Other): Adults (> 18 years of age)
  * Unilaterally implanted with an Advanced Bionics implant (CII or later)
  * At least six months of CI use experience
  * Limited bimodal benefit as perceived by the recipient and/or the clinician
  * Participants may or may not currently be using a hearing aid in the unimplanted ear.
  * Open set performance with current device configuration:
    * ≥40% AzBio sentence score in quiet (S0)
    * If currently bimodal:
  * Hearing aid ear only CNC score <50%
  * AzBio Scores bimodal benefit <15%
  * Unaided audiometric threshold of ≤100 dBHL up to 500 Hz
  * Ability and willingness to participate in multiple sets of open speech testing (and chronically evaluate HA and CROS benefit)
  Interventions: Device: Naida Hearing Aid; Device: Naida Contralateral Routing of Sound Device
- Naida CROS Device (Other): The same cohort will cross over to each arm.
  Interventions: Device: Naida Hearing Aid; Device: Naida Contralateral Routing of Sound Device

INTERVENTIONS:
Device: Naida Hearing Aid — hearing aid
  Other Names: HA
Device: Naida Contralateral Routing of Sound Device — This is a device that routes sound to the non-cochlear implanted ear.
  Other Names: CROS

SUMMARY:
The rationale is to determine (in individuals with limited perceived bimodal benefit) whether the CROS device may be a better solution for obtaining two-sided input. If yes, this study would be practice-changing.

DETAILED DESCRIPTION:
It is well accepted that bilateral input can significantly improve speech understanding in noise for patients with cochlear implants. For cochlear implant (CI) recipients who have a CI on only one side, two sided input can be provided with simultaneous use of a hearing aid (HA) or a CROS device on the opposite side. The decision about which device to use depends on the level of residual hearing a recipient has in non CI-implanted ear, and more specifically what level of useable residual hearing s/he has. Access to useable low frequency hearing can not only improve speech understanding in noise, it can also improve sound quality, pitch perception and music perception.

Clinicians can reasonably predict that a recipient with hearing thresholds better than 60 dB HL at low frequencies (below 750 Hz) would benefit from amplification. For recipients with no measurable acoustic hearing in the contralateral ear, CROS would be a reasonable option, especially if bilateral implantation is not feasible or desired. However, it is more difficult to predict the appropriate device in individuals who have some measurable acoustic hearing but may be receiving limited benefit from it. This can be especially challenging because audiometric thresholds are not a reliable predictor of bimodal benefit. Additionally, acoustic hearing can provide subjective benefits which could hold different intrinsic value or significance for different individuals depending on their life style and listening needs.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years of age)
* Unilaterally implanted with an Advanced Bionics implant (CII or later)
* At least six months of CI use
* Limited bimodal benefit as perceived by the recipient and/or the clinician
* Participants may or may not currently be using a hearing aid in the unimplanted ear.
* Open set performance with current device configuration:
* ≥40% AzBio sentence score in quiet (S0) and? (i.e. do both these apply)

If currently bimodal:

* Hearing aid ear only CNC score <50%
* AzBio Scores bimodal benefit <15% increase in score compared to CI only?
* Unaided audiometric threshold of ≤100 dBHL up to 500 Hz
* Ability and willingness to participate in multiple sets of open speech testing (and ongoing evaluation of HA and CROS benefit)

Exclusion Criteria:

* Patients who are not proficient in English as the AzBio testing is available in English only.
* Patients with agenesis of the contralateral ear

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-03-20 (Estimated)

PRIMARY OUTCOMES:
Perception of speech by way of audiogram and AzBio word testing. | At Baseline, Week 6 and Week 12
  Change in perception of speech by way of audiogram (hearing threshold across dB and frequencies) and AzBio word testing (% accuracy).
7 point Likert study-specific scales illuminating subjective feedback of experience using HA or CROS | At Baseline, Week 6 and Week 12
  Change in 7 point Likert study-specific scales illuminating subjective feedback of experience using HA or CROS. 1 (very dissatisfied) to 7 (very satisfied)
Participant narrative illuminating subjective feedback of experience using HA or CROS | At Baseline, Week 6 and Week 12
  Evolution of narrative interview themes illuminating subjective feedback of experience using HA or CROS

SECONDARY OUTCOMES:
Demographics | At Baseline
  Age, Gender, Hearing History

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, ON - Ontario, Canada

IPD SHARING:
Plan to Share IPD: No